CLINICAL TRIAL: NCT00259142
Title: Community Acceptability and Cost-effectiveness of Two Drug Distribution Methods for Home Based Management of Fevr in Kayunga District, Uganda
Brief Title: Acceptability and Cost Effectiveness of Home Based Management of Fever: Different Strategies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started
Sponsor: DBL -Institute for Health Research and Development (Other)
Collaborators: World Health Organization (Other); Institute for Epidemiology and Social Medicine, Aarhus University, Denmark (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UGA.5.2RNA2005
Record Dates: First submitted 2005-11-25; First posted 2005-11-29 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Fever; Anaemia; Malaria
Keywords: home management of fever, malaria, Uganda
MeSH Terms: conditions — Fever; Anemia; Malaria | interventions — Chloroquine; fanasil, pyrimethamine drug combination

INTERVENTIONS:
Drug: Chloroquine, sulphadoxine-pyrimethamine

SUMMARY:
Malaria remains a major cause of morbidity and mortality particularly among children < 5 years in Uganda. Due to inaccessibility many children die before they reach the health facility. The Home Based Management of Fever (HBMF) strategy was adopted in Uganda as a mean to improve access to early and appropriate treatment of fever at community level. Pre-packed chloroquine with sulphadoxine-pyrimethamine (HOMAPAK) is provided through Community Drug Distributors(CDDs). Initial evaluation showed underutilization of the CDDs (15%). This cast doubt on community acceptability, accessibility as well as its feasibility and cost effectiveness. This 3-year project intends to compare community acceptability and cost effectiveness of two HOMAPAK distribution methods. The current CDD-based HOMAPAK distribution versus home-based HOMAPAK distribution. The study hypothesis is that "home-based HOMAPAK distribution is more acceptable to the community and more cost effective than the CDD based HOMAPAK A non randomised community study will be conducted in two sub-counties of Mukono district. In the control arm, HOMAPAKs will be distributed through the CDDs while in the intervention arm, HOMAPAKs will be directly distributed to the caretakers in the homes. The study population are caretakers and their children < 5 years. At baseline a survey (Phase 1) with a sample size 657 in each study area will assess the common drugs stocked at home to treat malaria and the health seeking behaviour for malaria for children < 5 years and to determine the prevalence of malaria parasitaemia and anaemia among children < 5 years. Phase 2 includes the intervention. The villages will be assigned to either the control or intervention arm. Anaemia and malaria parasitaemia among children with fever will be assessed through active case finding. The impact of either distribution system on accessibility, acceptability, sustainability, compliance, cost effectiveness and malaria morbidity will be assessed during the evaluation phase. Health education messages on malaria prevention and treatment will be given to both communities. Drug misuse will be limited by distributing HOMAPAKs according to the number of children <5years in each household. HOMAPAK will only be replenished after the caretaker returns a used packet to the CDD.

DETAILED DESCRIPTION:
The hypothesis is that distributing HOMAPAK directly to caretakers is more acceptable to the community, cost effective and results in reduced malaria morbidity among children < 5 years than distribution through CDDs.

General Objective:

To compare the communities malaria seeking behaviour in the two drug distribution methods of HOMAPAK in order to provide information that can be used to enhance the HBMF strategy.

Specific Objectives:

1. To assess trends in the types and numbers of antimalarials stocked for use among children < 5 years in the two study areas
2. To assess the patterns of health seeking behaviour in the community for fever among children under five years of age.
3. To assess the incidence of malaria, and the associated morbidity (anaemia) in the two study areas.
4. To compare community acceptability of the two drug distribution methods of HOMAPAK in the aspects of, utilisation of the services, drug compliance, coverage and accessibility.
5. To assess the cost and compare cost effectiveness of the two drug distribution methods of the HOMAPAK on malaria morbidity in the community.

   Study area and population:

   The study will be conducted in Kayunga district, located 80 km northeast of Kampala with a total population of 800000 (Uganda Housing and Population Census, 2002) of which 20 % is < 5 years. It is hyperendemic for malaria. The study population will consist of the children < 5 years and their caretakers. The study areas will be those without HOMAPAK being distributed at all.

   Study design:

   Household based intervention study. Two drug distribution methods of HOMAPAK will be compared. In the Control arm, HOMAPAKs will be distributed through the conventional HOMAPAK distribution method (i.e through the CDDs) while in the Intervention arm, HOMAPAKs will be distributed directly to the caretakers.

   A Baseline survey will assess the patterns of health seeking behaviour for the < 5 children with fever. Types of antimalarials stocked in homes will be established. The prevalence of malaria and anaemia among children < 5 years will be established. In the intervention phase the two different HOMAPAK distribution methods will be implemented and monitored. Active case finding of malaria cases will be combined with passive surveillance. A structured questionnaire will be administered to the caretakers and a finger prick blood sample for Hb and malaria parasitaemia will be drawn from the children. Malaria records at the health facility will be reviewed for number of malaria cases seen and their clinical outcome. In the evaluation phase the impact of the drug distribution methods on antimalarials stocked in the homes,health seeking behaviour and other outcome measures.

   Sample size:

   Baseline and evaluation phase The sample size (n) has been estimated according to Kirkwood and Sterne (2003) for comparing of two means. The required sample size is 597 per group. To cater for loss of follow up, 10 % of the sample size will be added thus giving a total of 657 per group.

   Methods The Intervention Phase The study populations will consist of the caretakers and children under five years of age in the Control and the Intervention arms. Two CDDs in each village will be trained and given HOMAPAKs. In the Control Arm the CDDs will keep the HOMAPAKs and will only be distributed when the caretakers seek care for their children. In contrast in the intervention area, the CDDs will distribute the drugs to all homes with children < 5 years of age. The CDDs will only act as RELAY POINTS for the HOMAPAKs. All villages of the study parishes in either arm will be included.

   Activities:

   Community sensitisation/selection of the CDDs Through village meetings the community will be informed about the project and be requested to select two people for training as CDDs. Two district trainers will conduct a training workshop. Item included: the roles of the CDD, issues about malaria (its importance, cause, clinical presentation, case management & prevention), HOMAPAK dosage, counselling (preventive, compliance), referral of cases, record keeping (HMIS, drug stocks), recognition of a child with fever and what to do for her/him, determining what pre-pack to give, recording the treatment and drug storage.

   Procurement and distribution of HOMAPAK HOMAPAKs will be procured through the MoH and supplied to all CDDs in both study communities. The CDDs in the control arm will only give the drugs when the caretakers seek care, while those in intervention arm will distribute the appropriate HOMAPAKs to all HH with children < 5 years. In order to prevent drug misuse, the CDDs in the intervention group will be instructed to only replenish the stocks in the household after the caretaker produces the used packet of HOMAPAK.

   Monitoring cases of malaria Three field assistants (FAs) will be stationed in the community and will do weekly surveys in households with children with either malaria or history of fever in the previous 7 days. A case of malaria will be any child, who either currently has a fever (axillary temperature >37.5 C) and any parasitaemia) or has a history of fever in 48 hours prior to the survey plus any parasitaemia. Information regarding health-seeking behaviour by the caretaker for the child with fever and related costs will be obtained by use of a questionnaire. Finger prick blood samples for Hb and malaria parasitaemia will be taken from the child. The Hb will be obtained by use of a portable haemoglobin photometer (HemoCue) while a thick malaria slide will be examined under a microscope. The FAs will give appropriate information regarding malaria control and treatment to the caretakers.

   Monitoring and Supervision of project activities Project activities will be monitored and supervised by the project staff , the district health team, and the community themselves. The project staff will join the district team during their quarterly support supervision visits. The PI and the district supervisor will do fortnightly supervision in the study area. During the supervisory visits, meetings with the CDDs and community leaders will be held to discuss the progress of the project activities. Meetings will also be held with the FAs and Field Supervisors. Patient records and drug stock cards at both the health facility and CDDs will be reviewed.

   The Evaluation Phase:

   To assess the impact of the distribution methods on patterns of health seeking behaviour of the caretakers for fever among children < 5 years, acceptability and related costs for the household and government, antimalarials stocked in the homes, malaria morbidity among children < 5 years, a second KAP Survey will be conducted 2 years after the implementation of the project, in the same villages, on a comparable sample of 657 caretakers and children < 5 years in each study area using the same structured questionnaire and FGD guide.

   Sampling:

   Two sub counties (SC) in the district with similar demographic and socio-economic characteristics will be purposely selected. 50% of the parishes in each SC will then be randomly selected.

   Baseline and Evaluation phase:

   In order to have at least 30 households (HH) in a village, a total of 17 villages will be selected from the sampled parishes in each sub county using probability proportionate to size sampling. At village level the list of all the HH in the village will be obtained from the chairman of the village. The 30HH will be selected randomly. Appointments will be made with the caretakers to agree on the time for the interview. In case the caretakers refuse to participate, she will not be replaced. In case the selected HH does not have a child < 5 years, it will be replaced by one in the neighbourhood with such a child. In case there is more than one eligible caretaker in the selected HH like in polygamous homes, then one respondent will be selected by use of the ballot method. A similar procedure will be applied in case there is more than one eligible child in the HH. After seeking an informed consent from the respondent, an interview will be conducted.Participants for the FGDs will be purposely selected from the parishes HH that will not be part of the structured questionnaire. Two FGDs for men and Two for women will be conducted separately.

   Intervention phase:

   All households with children < 5 years in the study villages in both the control and intervention arm

   Outcome Measures:

   Patterns of health seeking behaviour
   * Types of health services used, factors affecting utilisation of the formal health services (individual, community, health system based etc)

   Utilisation of antimalarial in the community
   * Types of antimalarial drugs used for the malaria among the under five children
   * Number of antimalarial drugs used to treatment an episode of fever
   * % change in types and number of antimalarial drugs stocked in the homes

   Acceptability
   * Proportion of under-five children with fever that are given HOMAPAKS
   * Proportion of caretakers that use HOMAPAKS as their first choice of treatment for fever
   * Proportion of caretakers that are able to correctly use HOMAPAKs

   Accessibility

   - Proportion of children that get treatment with HOMAPAK within 24 hours of onset of fever
   * % of weeks in the year without stock-outs of HOMAPAKs
   * % of drug distributors that are always available
   * % of households with HOMAPAKS for future episodes of fever

   Feasibility/Sustainability

   - % of distributors/households with satisfactory drug storage,% of households with expired HOMAPAK

   Compliance
   * Proportion of febrile under-five children that get appropriate treatment
   * % of caretakers that show correct dosage for the child
   * % of under-five children that are given HOMAPAK for only fever/malaria
   * proportion of under five that get appropriate referral

   Coverage

   - Proportion of under five children with fever that get treatment with HOMAPAK

   Cost & cost-effectiveness

   - Average costs incurred by MoH to deliver HOMAPAK up to HH level

   - Average costs incurred by MoH in treatment of a severe malaria case in a health facility

   - Average Costs incurred by a house hold level to seek care for a case of malaria

   - Average cost by a household to treat a case of severe malaria at a health facility

   - Cost effective ratio for a case of severe malaria averted at health facility level

   - Cost effective ratio for a case of blood transfusion averted at health facility level

   Malaria morbidity
   * % increase in mean Hb levels
   * % decrease in prevalence and intensity of parasitaemia
   * % decrease in severe malaria cases (HIS)

ELIGIBILITY:
Inclusion Criteria:

* children 0-59 months with fever

Max Age: 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1314 (Estimated)
Dates: Start 2005-11; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
See detailed description

SECONDARY OUTCOMES:
See detailed description

CONTACTS AND LOCATIONS:
Overall Officials: Robinah Najjembe, MD, MPH, Principal Investigator — Makerere University Institute of Public Health
Locations (1):
- Kayunga District, Kayunga, Uganda

REFERENCES:
- See also: Related Info — http://www.dbl.life.ku.dk/